CLINICAL TRIAL: NCT05288543
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Food Effect of Orally Administered IPG7236 in Healthy Adult Participants
Brief Title: A Study of Orally Administered IPG7236 in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nanjing Immunophage Biotech Co., Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPG7236-A002
Record Dates: First submitted 2022-03-17; First posted 2022-03-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose Phase (Experimental): Drug: IPG7236 Dosage form: Tablet Route of Administration: Oral Dose level: Cohort 1 (25 mg), Cohort 2 (50 mg), Cohort 3 (100 mg), Cohort 4 (200 mg), Cohort 5 (300 mg), Cohort 6 (400 mg), Cohort 7 (500 mg) and Cohort 8 (600 mg)
  Interventions: Drug: IPG7236- Single ascending dose
- Multiple Ascending Dose Phase (Experimental): Drug: IPG7236 Dosage form: Tablet Route of Administration: Oral Dose level: Cohort 1 (100 mg), Cohort 2 (300 mg) and Cohort 3 (500 mg)
  Interventions: Drug: IPG7236- Multiple ascending dose
- Part A (Placebo) (Placebo Comparator): Placebo tablets identical to IPG7236 tablets Dosage form: Tablet Route of Administration: Oral
  Interventions: Other: Placebo (Part A)

INTERVENTIONS:
Drug: IPG7236- Single ascending dose — Subjects will receive IPG7236 tablets orally once on Day 1 in a fasted state
  Arms: Single Ascending Dose Phase
Drug: IPG7236- Multiple ascending dose — Subjects will receive IPG7236 tablets orally once daily for 10 days from Day1 to Day 10 in a fasted state
  Arms: Multiple Ascending Dose Phase
Other: Placebo (Part A) — Subjects will receive IPG7236 tablets orally once on Day 1 (Part A) or once daily for 10 days from Day1 to Day 10 (Part B) in a fasted state
  Arms: Part A (Placebo)

SUMMARY:
The study is a phase 1, randomized, double-blind, placebo-controlled, single and multiple dose escalation study to evaluate the safety, tolerability, pharmacokinetic and food effect of orally administered IPG7236 in healthy adult participants.

DETAILED DESCRIPTION:
The study consists of two parts

Part A (Single ascending dose): There are total 8 Single Ascending Dose cohorts.

Dose levels are as follows Cohort 1: 25 mg of IPG7236 or placebo as per the randomization code, Cohort 2: 50 mg of IPG7236 or placebo as per the randomization code Cohort 3: 100 mg of IPG7236 or placebo as per the randomization code Cohort 4: 200 mg of IPG7236 or placebo as per the randomization code Cohort 5: 300 mg of IPG7236 or placebo as per the randomization code Cohort 6: 400 mg of IPG7236 or placebo as per the randomization code Cohort 7: 500 mg of IPG7236 or placebo as per the randomization code Cohort 8: 600 mg of IPG7236 or placebo as per the randomization code In Cohort 1 total of 6 subjects enrolled. The 4 subjects will receive IPG7236 and 2 subjects will receive the placebo as per the randomization code.

In Cohort 2 to Cohort 8, 6 subjects will receive IPG7236 and 2 subjects will receive the placebo as per the randomization code.

Part B (Multiple ascending dose): There are total 3 Multiple ascending dose cohorts.

Dose levels are as follows Cohort 1: 100 mg of IPG7236 or placebo as per the randomization code Cohort 2: 300 mg of IPG7236 or placebo as per the randomization code Cohort 3: 500 mg of IPG7236 or placebo as per the randomization code Total of 8 subjects per cohort, 6 subjects will receive IPG7236 and 2 subjects will receive placebo per the randomization code The Multiple Ascending Dose phase of Cohort 1, Cohort 2 and Cohort 3 will commence based on the safety and tolerability data obtained from Single Ascending Dose phase of Cohort 4, Cohort 6 and Cohort 8.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female participants between 18 and 55 years of age (inclusive).
2. Body weight between 45 and 100 kg (inclusive) and body mass index (BMI) within 18~32 kg/m2 (inclusive).

   Health status
3. In good health as determined by screening tests. Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, full physical examination (including measurement of blood pressure and pulse rate), 12-lead Electrocardiograph (ECG), and clinical laboratory tests.

   * Vital signs (measured after resting for 5 minutes semi-supine position) within a normal range of the clinical site,, or outside the normal range and not considered clinically significant by the Investigator.
   * Standard 12-lead Electrocardiograph (ECG) parameters (recorded after resting for 5 minutes in semi-supine position) in the following ranges; QTc (Fridericia algorithm recommended) ≤ 450 ms for males and 470 ms for females, and normal ECG tracing, or abnormal ECG tracing not considered clinically relevant by the Investigator.
   * Laboratory parameters demonstrating no clinically significant abnormalities, as determined by the Investigator. Total bilirubin outside the normal range may be acceptable if total bilirubin does not exceed 1.5x ULN with normal conjugated bilirubin (with the exception of a patient with documented Gilbert syndrome).
4. A negative result on urine drug screen and a repeat negative result on Day -1 (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
5. Female participants must not be pregnant or breastfeeding and must use an effective contraception method with the exception of participants who have undergone sterilization more than 3 months prior to screening or who are postmenopausal.

   A woman of childbearing potential (WOCBP) must undergo pregnancy testing prior to the first dose of the study drug. The participant must be excluded from the study if the serum pregnancy test is positive.

   A postmenopausal state is defined as 12 months of amenorrhea without an alternative medical cause. In the absence of 12 months of amenorrhea, menopause may be confirmed by follicle stimulating hormone (FSH) measurement (> 40 IU/L or mIU/mL).

   Females on HRT (Hormonal Replacement therapy), where menopausal status is indeterminate, will be required to use a non-estrogen hormonal contraceptive method if participants wish to continue their HRT during the study. Participants must otherwise discontinue HRT to allow for confirmation of postmenopausal status prior to enrollment in the study.
6. Provide written informed consent prior to undertaking any study-related procedures.
7. Must not be under any administrative or legal supervision or under institutionalization as per a regulatory or juridical order.

Exclusion Criteria:

1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, musculoskeletal, rheumatological, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
2. Frequent severe headaches and/or migraines, recurrent nausea and/or vomiting (defined as vomiting more than twice a month).
3. Made a blood or plasma donation of ≥500 ml within 1 month prior to the first dose.
4. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions, which in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
5. Known hypersensitivity to any component of the IMP formulation.
6. History or presence of drug or alcohol abuse (defined as alcohol consumption of more than 2 units per day on a regular basis).
7. Regular smoking (defined as more than 5 cigarettes or equivalent per week), or unable to stop smoking during the study. Occasional smokers may be enrolled but need to abstain during admission to the site
8. Excessive consumption of beverages containing xanthine bases (defined as more than 4 glasses per day).
9. Any medication, including St John's Wort, within 14 days prior to administration of the first dose or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception, menopausal hormone replacement therapy, or occasional paracetamol at doses up to 2g/day.
10. Any consumption of grapefruit or products containing grapefruit within 5 days prior to the first dose administration.
11. Any vaccination in the 2 weeks prior to administration of the first dose (Covid19 vaccination included, and planned COVID19 vaccinations, including booster shots, during the study or for 2 weeks after the last dose of the study drug)
12. Any participant who, in the judgment of the Investigator, is likely to be non-compliant during the study, or to be unable to cooperate due to language problems or poor mental development.
13. Any participant who enrolled in or participated in any other clinical study involving an investigational medicinal product, or in any other type of medical research within 1 month or within 5 times the elimination half-life prior to administration of the first dose.
14. Any participant who cannot be contacted in the case of an emergency.
15. Any participant who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof directly involved in conducting the study or any person dependent on (employees or immediate family members) the study site, the Investigator or the Sponsor.

    Biological status
16. Positive result on any of the following tests: hepatitis B surface antigen (HbsAg), hepatitis B core antibodies (HbcAb), anti-hepatitis C virus antibodies (anti-HCV), anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
17. Positive alcohol test at D-1.
18. Any participant in whom venous blood collection is difficult.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of IPG7236 after ascending single oral doses through adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events v5 | Up to 36 days
To assess the safety and tolerability of IPG7236 after ascending multiple oral doses through adverse events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events v5 | Up to 45 days

SECONDARY OUTCOMES:
To assess the pharmacokinetic (PK) parameters of IPG7236 after ascending single oral doses | Up to 36 days
  Plasma PK parameters: Cmax (maximum plasma concentration)
To assess the pharmacokinetic (PK) parameters of IPG7236 after ascending single oral doses | Up to 36 days
  Plasma PK parameters: Tmax (time to Cmax)
To assess the pharmacokinetic (PK) parameters of IPG7236 after ascending multiple oral doses | Up to 45 days
  Plasma PK parameters: Css,max (maximum plasma concentration at steady state)
To assess the pharmacokinetic (PK) parameters of IPG7236 after ascending multiple oral doses | Up to 45 days
  Plasma PK parameters: CTss,max (time to maximum plasma concentration at steady state)
To evaluate the effect of food on the PK of IPG7236 | Up to 45 days
  Pharmacokinetics parameters using Cmax (maximum plasma concentration)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia